CLINICAL TRIAL: NCT00751439
Title: Verification of Pulse Oximetry in Neonatal Population
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Mark Mammel, M.D., Children's Hospitals & Clinics of Minnesota
Other Study IDs: 0802-024
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Respiratory Distress Syndrome
Keywords: Oximeter; Arterial blood gas; comparison
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this his post-market, observational study titled Verification of Pulse Oximetry in the Neonatal Population is to gather data to further support the accuracy of Nonin's pulse oximeters when used in the neonate population. Neonates who are currently undergoing arterial blood gas (ABG) sampling, as part of their medical care will be recruited to participate in this study for collecting opportunity samples. Nonin's PureLight® noninvasive sensor will be applied to a foot of the neonate; an adhesive wrap secures the sensor to the neonate. The sensor immediately begins obtaining SpO2 and pulse rate measurements which are sent to the oximeter module for display on the Electronic Data Collection System (EDCS). At the time the prescribed ABG is drawn, the EDCS must have a marker captured to identify the end of the ABG for SpO2 comparison. The SpO2 accuracy of pulse oximeter will be measured by comparing SpO2 readings of the pulse oximeter to values of SaO2 (opportunity samples) determined by a CO-oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 25 weeks to full term
* Weight range: No minimum or maximum range
* Age: up to 1 month (30 DAYS)
* Gender: Both
* ABGs as part of their medical care, to be analyzed by co-oximeter
* Consent signed by at least one legal guardian

Exclusion Criteria:

* Presence of any skin irritation or breakdown on the foot
* Foot impediments which would preclude proper placement of the sensor
* Clinical condition precluding the use of adhesive materials
* Cessation of ABGs during study enrollment

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates 25 weeks gestation to full term
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Mammel, M.D., Principal Investigator — Children's Hospitals & Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States